CLINICAL TRIAL: NCT06015386
Title: Clear Aligner Versus Removable Inclined Plane in Treatment of Anterior Crossbite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Salah, teaching assistant, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACB
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Anterior Crossbite
Keywords: clear aligner , anterior crossbite , inclined plane
MeSH Terms: interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inclined plane (Experimental): group treated with inclined plane
  Interventions: Other: inclined plane
- clear aligner (Experimental): group treated with clear aligner
  Interventions: Other: clear aligner

INTERVENTIONS:
Other: inclined plane — 2 parallel groups one treated with clear aligner and other treated using inclined plane
  Arms: inclined plane
Other: clear aligner — 2 parallel groups one treated with clear aligner and other treated using inclined plane
  Arms: clear aligner

SUMMARY:
the study is carried in faculty of dentistry Mansoura university to compare the efficiency and health quality life improvement between clear aligner and inclined plane in treatment of anterior crossbite

DETAILED DESCRIPTION:
the study *include 24 patient each group include 12 patient where randomly allocated and intra-oral scanning is done for them followed by software designing ,printing using PETG sheets of 0.75 in aligner group while in inclined plane the appliance is formed in conventional way.

ELIGIBILITY:
Inclusion Criteria:1. Patients age (7-12) years. 2. anterior crossbite 3. More than one tooth in a crossbite. 4. Favorable oral hygiene 5. No oral habits 6. ANB within the normal range i.e. (The crossbite will be diagnosed as functional or dental)

-

Exclusion Criteria:

1. Systemic conditions that may interfere with the treatment.
2. Bad habits that might jeopardize the appliance.
3. Transverse discrepancy.
4. Previous orthodontic treatment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
(OHRQoL (Oral Health-related Quality of Life) | 4 month
  CPQ8-10 scores at two different points in time.

SECONDARY OUTCOMES:
cephalometric analysis of data | 4 month
  compare cephalometric variables between two groups
3D model measurements | 4 month
  compare 3D model measurements variable between 2 group

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salem AS, Albelasy NF, El-Bialy AA. Effectiveness of clear aligner versus removable inclined plane in treatment of anterior crossbite in mixed dentition: A randomized clinical trial. J World Fed Orthod. 2025 Jun;14(3):125-130. doi: 10.1016/j.ejwf.2024.11.001. Epub 2024 Dec 19. PMID 39706691